CLINICAL TRIAL: NCT03203915
Title: Metabolic Response to Chardonnay Grape Marc Powder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: Sonomaceuticals LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 81946-4
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Dyslipidemia; Obesity
Keywords: cholesterol; triglyceride; grape seed extract; chardonnay marc powder; polyphenol; gut microbiome
MeSH Terms: conditions — Dyslipidemias; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): Order of treatments:
  A: Chardonnay grape marc powder high polyphenol dose B: Chardonnay grape marc powder low polyphenol dose C: Placebo
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)
- Group 2 (Experimental): Order of treatments:
  A: Chardonnay grape marc powder high polyphenol dose C: Placebo B: Chardonnay grape marc powder low polyphenol dose
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)
- Group 3 (Experimental): Order of treatments:
  B: Chardonnay grape marc powder low polyphenol dose C: Placebo A: Chardonnay grape marc powder high polyphenol dose
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)
- Group 4 (Experimental): Order of treatments:
  B: Chardonnay grape marc powder low polyphenol dose A: Chardonnay grape marc powder high polyphenol dose C: Placebo
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)
- Group 5 (Experimental): Order of treatments:
  C: Placebo A: Chardonnay grape marc powder high polyphenol dose B: Chardonnay grape marc powder low polyphenol dose
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)
- Group 6 (Experimental): Order of treatments:
  C: Placebo B: Chardonnay grape marc powder low polyphenol dose A: Chardonnay grape marc powder high polyphenol dose
  Interventions: Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg); Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg); Dietary Supplement: Placebo (0mg)

INTERVENTIONS:
Dietary Supplement: Chardonnay grape marc marc high polyphenol dose (120mg) — 3 prepackaged capsules taken once in the morning with meal for 3 weeks. The total dose will be 120mg of total polyphenols
Dietary Supplement: Chardonnay grape marc powder low polyphenol dose (75mg) — 3 prepackaged capsules taken once in the morning with meal for 3 weeks. The total dose will be 75mg of total polyphenols
Dietary Supplement: Placebo (0mg) — 3 prepackaged capsules taken once in the morning with meal for 3 weeks. The total dose will be 0mg of polyphenols

SUMMARY:
To determine if the addition of chardonnay grape marc (also called pomace) powder enriched with grape seed extract to the diet will result in reducing blood levels of cholesterol or triglycerides.

DETAILED DESCRIPTION:
Previous research on grape seed nutritional properties has predominantly been confined to grape seed extracts (GSE) containing only soluble components. In animal models, GSE has been shown to prevent increases in blood pressure, blood cholesterol, and insulin resistance. In humans, there have been improvements in blood pressure, however no significant effect on blood cholesterol levels. Whole milled grape marc flours deliver more dietary complexity than seed extracts alone. In addition to the extractable and non-extractable polyphenols, flour offers dietary fiber, minerals, sterols and polyunsaturated fats. Grape marc flour is currently used as a food ingredient that is incorporated into various baked goods. However, to obtain good control of the dose level, the product will be provided in capsule form for this study. For reference, a ½ cup of of a high polyphenol food such as blueberries, contains about 325 milligrams of polyphenols, thus even with the higher dose, participants will be receiving an amount of polyphenols that is less than ¼ cup of blueberries. The grape marc powder is prepared in a facility that is certified for producing food-grade products, and the nutritional composition and safety of the product will be thoroughly evaluated before we begin the study. The objective of the current study is to determine if this chardonnay grape marc powder enriched with grape seed extract supplementation has beneficial impacts on the human blood lipid profile and to correlate gut biome changes to human metabolism.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25 and < 40 kg/m2
* Dyslipidemia as defined as (any one or all of the following values):
* Total cholesterol > 190 mg/dL but < 240 mg/dL
* LDL-cholesterol > 130 mg/dL but < 160 mg/dL
* HDL-cholesterol < 40 mg/dL (men)/<50 mg/dL (women)
* Fasting triglycerides > 150 mg/dL but < 300 mg/dL

Exclusion Criteria:

* Renal, cardiovascular, gastrointestinal or hepatic disease, by medical history
* History of a previous cardiovascular event
* Diagnosis of type 2 diabetes
* Pregnancy or lactation
* Use of tobacco
* Food sensitivities or allergies to the foods or components of foods provided in the standard meals including gluten, dairy, egg, soy, nuts, or seafood
* Use of herbal or plant-based supplements; omega-3 fatty acids, and fish oils in the past 3-6 months, and unwilling to discontinue use while participating in the study.
* Use of lipid-lowering, glucose-lowering, anti-hypertensive, or weight loss medications
* Use of antibiotics in the last three months.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Changes in lipid profile | Weeks 4, 10, 16
  Fasting triglyceride concentrations, LDL cholesterol, HDL cholesterol, non-HDL cholesterol will be measured in serum; postprandial triglyceride measurements (1, 2, 3 hours)

SECONDARY OUTCOMES:
Changes in fecal microbiome profile | Weeks 1, 4, 10, 16
  Gut microbiota community profile will be determined by 6M read metagenomic gene sequencing from stool samples
Changes in gut fermentation profile | Weeks 4, 10, 16
  Hydrogen and methane gas (parts per million) will be measured simultaneously in breath to assess gut fermentation
Changes in inflammatory markers | Weeks 4, 10, 16
  Immunological markers such as: tumor necrosis factor-α, Interleukin-β, Interleukin-6, Interleukin-1B, Interleukin-10, Interleukin-18, Interleukin-1a, Intercellular Adhesion Molecule 1, vascular cell adhesion molecule 1, C-reactive protein, Serum amyloid A, neopterin, myeloperoxidase, eotaxin, Interferon gamma-induced protein 10, Myeloid dendritic cell, monocyte chemoattractant protein 1, Matrix metalloproteinase-1, Matrix metalloproteinase-3, Matrix metalloproteinase-9 will be taken at fasting at each test day.
Changes in endothelial function measurement and blood pressure | Weeks 4, 10, 16
  Blood pressure will be measured each test day. Endothelial function will be measured once per day using peripheral arterial tone (PAT) signal technology. Endothelial function is expressed as a Reactive Hyperemia Index (RHI).
Changes in metabolomic profile | Weeks 1, 4, 10, 16
  Fecal bile acids, plasma bile acids, fecal and plasma short-chain fatty acids
  Fecal samples were taken at baseline and after each test day. Plasma samples were taken at fasting, 1, 2, and 3hrs postprandially.
Changes in cognitive function | Weeks 4, 10, 16
  Executive function will be assessed using Cambridge Neuropsychological Test Automated Battery (CANTAB) and Autonomic Nervous System Output.

OTHER OUTCOMES:
Changes in glucose metabolism | Weeks 4, 10, 16
  Glucose and insulin measures at fasting and postprandially (1, 2, 3 hrs). this includes assessing insulin resistance and sensitivity indexes using fasting measurements.
Changes in appetite hormones | Weeks 4, 10, 16
  Leptin, Ghrelin, Peptide YY 3-36, Glucagon-like peptide-1 at fasting and postprandial (1, 2, 3 hr)
Changes in body composition and energy expenditure | Weeks 4, 10, 16
  Body composition by Dual energy X-ray Absorptiometry scan (radiologic exposure), body weight, waist and hip circumference, indirect calorimetry measured each visit.
Changes in self-report of hunger and mood | Weeks 4, 10, 16
  Subjective rating measures using a visual analog scale at fasting and every 20 mins postprandially./
Changes in NMR lipid particle profile | Weeks 4, 10, 16
  cholesterol species (e.g. VLDL, IDL, LDL, etc) identified and their particle sizes (e.g. small, medium, large) identified at fasting and 3hr postprandial
Changes in oxidized LDL | Weeks 4, 10, 16
  oxidized LDL measured at fasting and 1, 2, 3 hrs postprandial
Changes in apolipoprotein profile | Weeks 4, 10, 16
  Apo CIII, Apo B, Apo AI, Apo E measured at fasting and postprandial (1 and 3hr)
General health | Weeks 4, 10, 16
  General well being via questionnaire, comprehensive metabolic panel (at fasting), fatty liver index

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Keim, PhD, Principal Investigator — United States Department of Agriculture (USDA)
Locations (1):
- Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No